CLINICAL TRIAL: NCT04378179
Title: Recognition of Heart Failure With Micro Electro-Mechanical Sensors (REFLECS)
Status: Completed | Type: Observational
Sponsor: Francois Haddad (Other)
Collaborators: Precordior Ltd (Industry)
Responsible Party: Sponsor-Investigator, Francois Haddad, Clinical Professor Medicine - Med/Cardiovascular Medicine, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 55057
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure; Pulmonary Hypertension
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- HFpEF: HF patients with preserved ejection fraction (HFpEF)
- HFrEF: HF patients with reduced ejection fraction (HFrEF)
- PH: Patients with Pulmonary hypertension (PH)
- Control: Elective patients visiting hospital cardiology who are not diagnosed with either HFpEF or HFrHF or PH but meet other inclusion criteria and none of the exclusion criteria.
- Controls with suspected CAD: Elective patients visiting hospital cardiology who are not diagnosed with either HFpEF or HFrHF or PH but meet other inclusion criteria and none of the exclusion criteria, and may have a diagnosis of Coronary Artery Disease (CAD) or may be suspected to have CAD.

SUMMARY:
The study will test the ability a novel wearable sensor based on a smartphone app (Precordior CardioSignal app) in combination with a sensor device (Suunto Movesense sensor) to non-invasively measure cardiac motion and function.

DETAILED DESCRIPTION:
Heart Failure (HF) is a syndrome where the heart is unable to pump or fill adequately to meet the circulatory needs of the body. The main purpose of this study is to test the ability a novel wearable sensor based on a smartphone app (Precordior CardioSignal app) in combination with a sensor device (Suunto Movesense sensor) to non-invasively measure cardiac motion and function. The phone and sensor are positioned on the chest and echocardiography is used as a gold standard to assess cardiac mechanics including myocardial strain, cardiac torsion, diastolic filling characteristics, hemodynamics including pressure estimates and stroke volume.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Able to consent in English and follow study instructions
* Patients hospitalized or being seen in clinic with heart failure with a diagnosis of HFpEF, HFrEF or PH, as corresponding to each target patient group
* Control patients may include patients that are hospitalized without heart failure, and cardiology patients without heart failure who are seen in outpatient cardiology, who may have suspected CAD and are scheduled for CCTA.

Exclusion Criteria:

* Severe cardiac valvular heart disease
* Previous prosthetic cardiac valve
* Pericardial disease including constrictive pericarditis or moderate or large pericardial effusion
* Mechanical circulatory support (including ECMO, LVADs etc).
* Heart and/or lung transplant recipients
* Major adverse cardiovascular event or surgery within 6 weeks of planned study enrollment
* Patients with pacemaker that has over 1% of beats paced
* Pectus excavatum (severe)
* Pregnant women
* On Dialysis
* Exclude at the clinical discretion of the Principal Investigators
* Not possible to acquire echocardiography with sufficient quality

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting Stanford Hospital and Clinics
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2023-10-07 (Actual)

PRIMARY OUTCOMES:
Heart failure detection | Baseline to Day 2
  Test the ability of the Precordior sensor to detect heart failure with reduced ejection fraction, heart failure with preserved ejection fraction and pulmonary hypertension compared to control participants. An additional comparison will be made to individuals without signs, diagnosed, or suspected HF who will be undergoing CCTA due to suspected CAD.

SECONDARY OUTCOMES:
Detection of differences in myocardial mechanics between admission and discharge | up to 2 weeks (during admission) and 2 to 14 weeks (during follow-up visit).
  The ability of the Precordior sensor to detect differences in myocardial mechanics as defined my myocardial longitudinal strain, hemodynamics and torsion analysis from admission and discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Haddad, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haddad F, Saraste A, Santalahti KM, Pankaala M, Kaisti M, Kandolin R, Simonen P, Nammas W, Jafarian Dehkordi K, Koivisto T, Knuuti J, Mahaffey KW, Blomster JI. Smartphone-Based Recognition of Heart Failure by Means of Microelectromechanical Sensors. JACC Heart Fail. 2024 Jun;12(6):1030-1040. doi: 10.1016/j.jchf.2024.01.022. Epub 2024 Apr 3. PMID 38573263